CLINICAL TRIAL: NCT05250466
Title: A Comparative Study on the Efficacy of AI Temperature-controlled Radiofrequency Technology and Electrical Stimulation in the Treatment of Vulvar Leukoplakia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vulvar leukoplakia 2022
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-10

CONDITIONS: Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency group (Experimental): AI Temperature-controlled Radiofrequency Technology
  Interventions: Procedure: Radiofrequency technology
- Electrical stimulation group (Active Comparator): Electrical Stimulation
  Interventions: Procedure: Electrical stimulation

INTERVENTIONS:
Procedure: Radiofrequency technology — The vulva and vagina were routinely disinfected with iodophor, the negative plate was placed on the patient's waist and abdomen, and the vulva module was selected for treatment for 10 minutes per side, for a total of 20 minutes. Parameters: power 10-20W, temperature 38-42C°, once every 10 days, 5 times in total
  Arms: Radiofrequency group
Procedure: Electrical stimulation — Routine vulvovaginal disinfection with iodophor, vaginal probes are placed in channel A, electrode pads are placed in channels B\C\D respectively, the frequency of electrical stimulation (the most comfortable amount) is adjusted, 10 times is a course of treatment, and mild lesions are treated for 1-2 courses of treatment , 2 to 3 courses of treatment for moderate to severe lesions.
  Arms: Electrical stimulation group

SUMMARY:
The study was designed as a prospective, multicenter, randomized, open-label, parallel-controlled clinical trial. The study population was patients with vulvar leukoplakia, and compared the efficacy and safety of AI temperature-controlled radio frequency technology and electrical stimulation in the treatment of vulvar leukoplakia. According to the research purpose, the sample size was calculated and determined to be 120 cases, and they were randomly assigned to the observation group and the control group according to the ratio of 1:1, namely 60 cases in the radio frequency observation group and 60 cases in the electric stimulation control group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed by pathological examination, meeting the diagnostic criteria for leukoplakia;
2. 18 to 60 years old;
3. Agree to sign the informed consent;

Exclusion Criteria:

1. Patients with severe liver and kidney dysfunction;
2. Combined with HIV, syphilis infection, acute vaginitis, cervical cancer;
3. Patients with cardiovascular disease;
4. People with hematological diseases;
5. Patients with hypertension and diabetes;
6. People with mental illness;
7. Pregnant and lactating women.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy index | 6 month after treatment
  Efficacy index: (score before treatment-score after treatment)/(score before treatment)×100%

SECONDARY OUTCOMES:
Recurrence rate | 6 month after treatment
  Percentage of recurrence of genital itching 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuanzhen Zhang, Professor, Study Chair — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No